CLINICAL TRIAL: NCT00402831
Title: An Open, Randomised, Comparative, Multicentre Study of the Immunogenicity and Safety of ProQuad® When Administered by Intramuscular (IM) Route or Subcutaneous (SC) Route to Healthy Children Aged 12 to 18 Months
Brief Title: ProQuad® Intramuscular vs Subcutaneous
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V221-036; F05-MMRV-304 (Other: MCMVaccBV (SPMSD) Protocol Number); 2006-001986-40 (EudraCT Number)
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intramuscular ProQuad® (Experimental): Participants will receive doses of ProQuad® by IM injection on Day 1 and Day 30 into the deltoid muscle perpendicular to the skin, with the first dose in the right arm and the second dose in the left arm.
  Interventions: Biological: ProQuad®
- Subcutaneous ProQuad® (Active Comparator): Participants will receive doses of ProQuad® by SC injection on Day 1 and Day 30 in the deltoid area at a 45° angle to the skin, with the first dose in the right arm and second dose in the left arm.
  Interventions: Biological: ProQuad®

INTERVENTIONS:
Biological: ProQuad® — Each dose (0.5 mL) contains live attenuated versions of measles virus Enders' Edmonston strain, mumps virus Jeryl Lynn™ (Level B) strain, rubella virus Wistar RA 27/3 strain, and varicella virus Oka/Merck strain.

SUMMARY:
Primary objective:

To demonstrate that two doses of ProQuad® administered by IM route are as immunogenic as two doses of ProQuad® administered by SC route to healthy children 12 to 18 months of age in terms of antibody response rates to measles, mumps, rubella and to varicella at 42 days following the second dose of ProQuad®

Secondary objectives:

* To describe the antibody response rates to measles, mumps, rubella and varicella measured 30 days following the first dose of ProQuad® administered by IM or SC route,
* To describe the antibody titres to measles, mumps, rubella and varicella at 30 days following the first dose and at 42 days following the second dose of ProQuad® both administered by IM or SC route,
* To describe the safety profile of two doses of ProQuad® both administered by IM or SC route.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant of either gender,
* Age 12 to 18 months,
* Negative clinical history of measles, mumps, rubella, varicella and zoster,
* Consent form signed by both holders of the parental authority or by the legal representative
* Holder(s) of the the parental authority / legal representative able to understand the protocol requirements and to fill in the Diary Card.

Exclusion Criteria:

* Prior receipt of measles, mumps, rubella and/or varicella vaccine either alone or in any combination,
* Any recent (≤30 days) exposure to measles, mumps, rubella, varicella and/or zoster
* Any recent (≤3 days) history of febrile illness
* Any severe chronic disease,
* Active untreated tuberculosis,
* Known personal history of seizure disorder,
* Any known blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the haematopoietic and lymphatic systems,
* Any severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection,
* Any immune impairment or humoral/cellular deficiency, neoplastic disease or depressed immunity including those resulting from corticosteroid [any long-term (≥14 days) administration of systemic corticosteroid therapy given daily or on alternate days at high doses (≥2 mg/kg/day prednisone equivalent or ≥20 mg/day if weight more than 10 kg) within the previous 30 days] or other immunosuppressive therapy,
* Any previous (≤ 150 days) receipt of immune globulin or any blood-derived product or scheduled to be administered through Visit 3,
* Any recent (≤7 days) tuberculin test or scheduled tuberculin test through Visit 3,
* Any recent (≤30 days) receipt of an inactivated or a live vaccine or scheduled vaccination through Visit 3,

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 405 (Actual)
Dates: Start 2006-10-06 (Actual); Primary Completion 2007-05-11 (Actual); Study Completion 2007-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne FIQUET, MD, Study Director — SPMSD

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinicaltrials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Haas H, Richard P, Eymin C, Fiquet A, Kuter B, Soubeyrand B. Immunogenicity and safety of intramuscular versus subcutaneous administration of a combined measles, mumps, rubella, and varicella vaccine to children 12 to 18 months of age. Hum Vaccin Immunother. 2019;15(4):778-785. doi: 10.1080/21645515.2018.1549452. Epub 2019 Jan 8. PMID 30481110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 411 male and female participants (12 to 18 months of age) were selected for study entry at 33 sites in France. A total of 405 participants were randomized and received 2 doses of study drug.
Groups:
- Intramuscular ProQuad®: Participants received both doses (given on Day 1 and Week 4) of ProQuad® by IM injection into the deltoid muscle perpendicular to the skin, with the first dose in the right arm and the second dose in the left arm. Doses were separated by 30 to 44 days.
- Subcutaneous ProQuad®: Participants received both doses (given on Day 1 and Week 4) of ProQuad® by SC injection in the deltoid area at a 45° angle to the skin, with the first dose in the right arm and second dose in the left arm. Doses were separated by 30 to 44 days.
Period: Overall Study
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Started | 202 | 203
ProQuad® Dose 1 (Day 1) | 202 | 203
ProQuad® Dose 1 (Day 30) | 202 | 203
Completed | 201 | 200
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Non-compliance with protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad® | Total
Number analyzed (Participants) | 202 | 203 | 405
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.72 (1.44) | 13.65 (1.53) | 13.68 (1.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 94 | 199
  Male | 97 | 109 | 206

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Antibody Response Rate Criteria Six Weeks After Completing ProQuad® Treatment
Description: Antibody response rates were determined 6 weeks after the second dose of IM or SC ProQuad®. Measles, mumps and rubella antibody levels were determined using enzyme-linked immunosorbent assay (ELISA) and varicella antibody levels were determined with glycoprotein-based ELISA (gpELISA). Response rates were determined as follows: measles antibody titre ≥255 mIU/mL in participants with baseline titre <255 mIU/mL; mumps antibody titre ≥10 ELISA Ab units/mL in participants with baseline titre <10 ELISA Ab units mL; rubella antibody titre ≥10 IU/mL in participants with baseline titre <10 IU/mL; varicella antibody titre ≥5 gpELISA units/mL in participants with baseline titre <1.25 gpELISA units/mL.
Time Frame: Week 10 (6 weeks after Dose 2 on Week 4)
Population: Participants who were initially seronegative to measles, mumps, rubella or varicella and who had post-vaccination serology results were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 153 | 148
Percentage of participants
  Measles: number analyzed (Participants) | 153 | 147
  Measles | 100 [97.6 to 100] | 100 [97.5 to 100]
  Mumps: number analyzed (Participants) | 152 | 148
  Mumps | 99.3 [96.4 to 100] | 99.3 [96.3 to 100]
  Rubella: number analyzed (Participants) | 129 | 132
  Rubella | 100 [97.2 to 100] | 99.2 [95.9 to 100]
  Varicella: number analyzed (Participants) | 138 | 134
  Varicella | 100 [97.4 to 100] | 99.3 [95.9 to 100]
Statistical Analysis 1: Comparison: Intramuscular ProQuad® vs Subcutaneous ProQuad®; Measles difference; Test type: Non-Inferiority or Equivalence — Noninferiority was declared when the lower bounds of the 95% confidence interval (CI) of the group difference in response rates was greater than -10%; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-2.5 to 2.6]
Statistical Analysis 2: Comparison: Intramuscular ProQuad® vs Subcutaneous ProQuad®; Mumps difference; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-3.0 to 3.3]
Statistical Analysis 3: Comparison: Intramuscular ProQuad® vs Subcutaneous ProQuad®; Rubella difference; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-2.3 to 4.1]
Statistical Analysis 4: Comparison: Intramuscular ProQuad® vs Subcutaneous ProQuad®; Varicella; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-2.1 to 4.1]

2. Secondary Outcome: Percentage of Participants Meeting Antibody Response Rate Criteria Four Weeks After the First ProQuad® Dose
Description: Antibody response rates were determined 4 weeks after the first dose of IM or SC ProQuad®. Measles, mumps and rubella antibody levels were determined using ELISA and varicella antibody levels were determined with gpELISA. Response rates were determined as follows: measles antibody titre ≥255 mIU/mL in participants with baseline titre <255 mIU/mL; mumps antibody titre ≥10 ELISA Ab units/mL in participants with baseline titre <10 ELISA Ab units mL; rubella antibody titre ≥10 IU/mL in participants with baseline titre <10 IU/mL; varicella antibody titre ≥5 gpELISA units/mL in participants with baseline titre <1.25 gpELISA units/mL.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 153 | 149
Percentage of participants
  Measles: number analyzed (Participants) | 153 | 148
  Measles | 100 [97.6 to 100] | 97.3 [93.2 to 99.3]
  Mumps: number analyzed (Participants) | 152 | 149
  Mumps | 97.4 [93.4 to 99.3] | 91.3 [85.5 to 95.3]
  Rubella: number analyzed (Participants) | 129 | 133
  Rubella | 98.4 [94.5 to 99.8] | 100 [97.3 to 100]
  Varicella: number analyzed (Participants) | 138 | 136
  Varicella | 98.6 [94.9 to 99.8] | 98.5 [94.8 to 99.8]

3. Secondary Outcome: Antibody Geometric Mean Titres (GMT) to Measles Four Weeks After the First ProQuad® Dose
Description: Antibody titre levels to measles were determined 4 weeks after the first dose of IM or SC ProQuad®. Measles antibody levels were determined using ELISA. Titre levels were determined in participants with baseline measles titre <255 mIU/mL.
Time Frame: Week 4
Population: Participants who were initially seronegative to measles and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (mIU/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 153 | 148
Antibody titres (mIU/mL) | 4058.7 [3643.1 to 4521.8] | 3327.0 [2835.4 to 3903.9]

4. Secondary Outcome: Antibody GMT to Mumps Four Weeks After the First ProQuad® Dose
Description: Antibody titre levels to mumps were determined 4 weeks after the first dose of IM or SC ProQuad®. Mumps antibody levels were determined using ELISA. Titre levels were determined in participants with baseline mumps titres <10 ELISA Ab units mL.
Time Frame: Week 4
Population: Participants who were initially seronegative to mumps and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (ELISA Ab units/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 152 | 149
Antibody titres (ELISA Ab units/mL) | 120.0 [102.2 to 140.9] | 101.9 [84.2 to 123.2]

5. Secondary Outcome: Antibody GMT to Rubella Four Weeks After the First ProQuad® Dose
Description: Antibody titre levels to rubella were determined 4 weeks after the first dose of IM or SC ProQuad®. Rubella antibody levels were determined using ELISA. Titre levels were determined in participants with baseline rubella titre <10 IU/mL.
Time Frame: Week 4
Population: Participants who were initially seronegative to rubella and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (IU/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 129 | 133
Antibody titres (IU/mL) | 46.9 [39.7 to 55.4] | 50.9 [44.9 to 57.7]

6. Secondary Outcome: Antibody GMT to Varicella Four Weeks After the First ProQuad® Dose
Description: Antibody titre levels to varicella were determined 4 weeks after the first dose of IM or SC ProQuad®. Varicella antibody levels were determined with gpELISA. Titre levels were determined in participants with baseline varicella antibody titre <1.25 gpELISA units/mL.
Time Frame: Week 4
Population: Participants who were initially seronegative to varicella and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (gpELISA units/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 138 | 136
Antibody titres (gpELISA units/mL) | 25.0 [22.5 to 27.7] | 23.6 [20.9 to 26.7]

7. Secondary Outcome: Antibody GMT to Measles Six Weeks After Completing ProQuad® Treatment
Description: Antibody titre levels to measles were determined 6 weeks after the second dose of IM or SC ProQuad®. Measles antibody levels were determined using ELISA. Titre levels were determined in participants with baseline measles titre <255 mIU/mL.
Time Frame: Week 10 (6 weeks after Dose 2 on Week 4)
Population: Participants who were initially seronegative to measles and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (mIU/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 153 | 147
Antibody titres (mIU/mL) | 3953.7 [3497.2 to 4469.9] | 3748.6 [3270.9 to 4296.0]

8. Secondary Outcome: Antibody GMT to Mumps Six Weeks After Completing ProQuad® Treatment
Description: Antibody titre levels to mumps were determined 6 weeks after the second dose of IM or SC ProQuad®. Mumps antibody levels were determined using ELISA. Titre levels were determined in participants with baseline mumps titre <10 ELISA Ab units mL.
Time Frame: Week 10 (6 weeks after Dose 2 on Week 4)
Population: Participants who were initially seronegative to mumps and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (ELISA Ab units/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 152 | 148
Antibody titres (ELISA Ab units/mL) | 157.9 [138.6 to 180.0] | 168.8 [146.9 to 194.0]

9. Secondary Outcome: Antibody GMT to Rubella Six Weeks After Completing ProQuad® Treatment
Description: Antibody titre levels to rubella were determined 6 weeks after the second dose of IM or SC ProQuad®. Rubella antibody levels were determined using ELISA. Titre levels were determined in participants with baseline rubella titre <10 IU/mL.
Time Frame: Week 10 (6 weeks after Dose 2 on Week 4)
Population: Participants who were initially seronegative to rubella and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (IU/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 129 | 132
Antibody titres (IU/mL) | 92.8 [82.4 to 104.5] | 94.2 [83.2 to 106.6]

10. Secondary Outcome: Antibody GMT to Varicella Six Weeks After Completing ProQuad® Treatment
Description: Antibody titre levels to varicella were determined 6 weeks after the second dose of IM or SC ProQuad®. Varicella antibody levels were determined with gpELISA. Titre levels were determined in participants with baseline varicella antibody titre <1.25 gpELISA units/mL.
Time Frame: Week 10 (6 weeks after Dose 2 on Week 4)
Population: Participants who were initially seronegative to varicella and who had post-vaccination serology results were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titres (gpELISA units/mL)
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 138 | 134
Antibody titres (gpELISA units/mL) | 358.1 [300.1 to 427.4] | 261.8 [216.7 to 316.4]

11. Secondary Outcome: Percentage of Participants Experiencing an Injection-site Adverse Event (AE) or Vaccine-related Systemic AE After the First ProQuad® Dose
Description: An AE is any untoward medical occurrence in a participant administered an investigational medicinal product (IMP) and which does not necessarily have a causal relationship with the IMP. Injection-site AEs (e.g., erythema, swelling, pain) and systemic vaccine-related AEs (e.g., pyrexia) were AEs of interest.
Time Frame: From Day 0 up to Day 28 (up to 28 days after the first ProQuad® dose)
Population: All participants who received at least one dose of study drug and had safety follow-up data are included.
Measure: Number; unit: Percentage of participants
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 202 | 203
Percentage of participants
  Injection-site AEs | 17.8 | 28.6
  Vaccine-related systemic AEs | 8.9 | 8.4

12. Secondary Outcome: Percentage of Participants Experiencing an Injection-site AE or Vaccine-related Systemic AE After the Second ProQuad® Dose
Description: An AE is any untoward medical occurrence in a participant administered an IMP and which does not necessarily have a causal relationship with the IMP. Injection-site AEs (e.g., erythema, swelling, pain) and systemic vaccine-related AEs (e.g., pyrexia) were AEs of interest.
Time Frame: From Day 30 up to Day 58 (up to 28 days after the second ProQuad® dose)
Population: All participants who received at least one dose of study drug and had safety follow-up data are included.
Measure: Number; unit: Percentage of participants
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 201 | 200
Percentage of participants
  Injection-site AEs | 20.4 | 29.5
  Vaccine-related systemic AEs | 6.0 | 5.0

13. Secondary Outcome: Percentage of Participants Discontinuing From Study Therapy Due to an AE After the First ProQuad® Dose
Description: An AE is any untoward medical occurrence in a participant administered an IMP and which does not necessarily have a causal relationship with the IMP.
Time Frame: From Day 0 up to Day 28 (up to 28 days after the first ProQuad® dose)
Measure: Number; unit: Percentage of participants
Arm/Group | Intramuscular ProQuad® | Subcutaneous ProQuad®
Number analyzed (Participants) | 202 | 203
Percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 72 (AEs were monitored for 28 days after each dose, and Dose 2 could have been given up to 44 days after Dose 1).
Description: An AE is any untoward medical occurrence in a participant administered an investigational medicinal product (IMP) and which does not necessarily have a causal relationship with the IMP. Event data are presented separately for Dose 1 and Dose 2.
Groups:
- IM ProQuad® Arm: Dose 1: All participants who received the first dose of ProQuad® via IM injection are included.
- SC ProQuad® Arm: Dose 1: All participants who received the first dose of ProQuad® via SC injection are included.
- IM ProQuad® Arm: Dose 2: All participants who received the second dose of ProQuad® via IM injection are included.
- SC ProQuad® Arm: Dose 2: All participants who received the second dose of ProQuad® via SC injection are included.
Arm/Group | IM ProQuad® Arm: Dose 1 | SC ProQuad® Arm: Dose 1 | IM ProQuad® Arm: Dose 2 | SC ProQuad® Arm: Dose 2
Serious Adverse Events (participants affected / at risk) | 2/202 | 2/203 | 1/201 | 1/200
Other Adverse Events (participants affected / at risk) | 153/202 | 166/203 | 141/201 | 137/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM ProQuad® Arm: Dose 1 (N=202) | SC ProQuad® Arm: Dose 1 (N=203) | IM ProQuad® Arm: Dose 2 (N=201) | SC ProQuad® Arm: Dose 2 (N=200)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM ProQuad® Arm: Dose 1 (N=202) | SC ProQuad® Arm: Dose 1 (N=203) | IM ProQuad® Arm: Dose 2 (N=201) | SC ProQuad® Arm: Dose 2 (N=200)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 12 (14) | 7 (7) | 12 (12)
Teething (Gastrointestinal disorders) | 19 (21) | 17 (19) | 11 (12) | 12 (13)
Injection site erythema (General disorders) | 14 (14) | 40 (42) | 31 (31) | 54 (54)
Injection site pain (General disorders) | 23 (23) | 12 (12) | 20 (20) | 20 (20)
Pyrexia (General disorders) | 115 (158) | 125 (161) | 89 (124) | 82 (113)
Bronchitis (Infections and infestations) | 20 (20) | 16 (18) | 9 (9) | 12 (14)
Ear infection (Infections and infestations) | 22 (22) | 19 (20) | 21 (21) | 22 (24)
Nasopharyngitis (Infections and infestations) | 19 (19) | 18 (20) | 15 (15) | 17 (18)
Rhinitis (Infections and infestations) | 14 (15) | 13 (14) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (14) | 11 (11) | 7 (8)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 12 (12) | 25 (25)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 11 (11) | 10 (10)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 15 (16) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sanofi Pasteur MSD shall have sixty days to review these documents and may refuse to give its consent in part or whole for confidential reasons (including but not limited to intellectual property rights, whether patentable or not).